CLINICAL TRIAL: NCT01401621
Title: The Effect of a Scratch Off Prompt on Health Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 813606-1
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Blood Pressure Check (Hypertension Screening); Cholesterol Test (Lipid Disorder Screening)
Keywords: behavioral economics; nudge; scratch off; blood pressure check; cholesterol test

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Scratch-Off Test Name Condition (Experimental): The name of the test the recipient needs is hidden behind a scratchoff on the reminder
  Interventions: Behavioral: Scratchoff Prompt: Name of Test
- Scratch-Off Call to Action Condition (Experimental): The recipient will be prompted to scratch-off the paper in order to find out how to follow the recommendation that the test be received.
  Interventions: Behavioral: Scratchoff Prompt: Call to Action
- Control Condition (Experimental): A control condition with no scratch-off element.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Scratchoff Prompt: Name of Test — A prompt will have the recipient scratch off the message that reveals the name of the test that the recipient needs
  Arms: Scratch-Off Test Name Condition
Behavioral: Scratchoff Prompt: Call to Action — A prompt will have the recipient scratch off the message to find out how to follow the recommendation that the test be received.
  Arms: Scratch-Off Call to Action Condition
Behavioral: Control — No scratch-off element
  Arms: Control Condition

SUMMARY:
The goal of this project is to determine whether prompting the recipient of a health reminder mailing to scratch off targeted area.

DETAILED DESCRIPTION:
The investigators will randomly assign individuals with different scratch off messages to 3 groups. The investigators are interested in whether the scratch off message will result in an increase in compliance with the recommended health behavior.

ELIGIBILITY:
Inclusion Criteria:

* Indications according to Spring 2011 CDC criteria for a blood pressure check
* Indications according to Spring 2011 CDC criteria for a cholesterol test
* Employee at partner corporation that implemented the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84953 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants that schedule an appointment for receipt of the relevant test | up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Milkman, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States